CLINICAL TRIAL: NCT01810991
Title: Investigation of Hyperhidrosis Treatment Using the Nd: YAG 1440nm Wavelength Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN12-1440-BK-HID1
Record Dates: First submitted 2012-12-06; First posted 2013-03-14 (Estimated); Results first posted 2020-12-10 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: HYPERHIDROSIS
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nd:YAG Laser (Experimental): Nd:YAG 1440nm Laser
  Interventions: Device: Nd:YAG Laser

INTERVENTIONS:
Device: Nd:YAG Laser — Nd:YAG 1440nm Laser

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Nd:YAG 1440 nm wavelength laser for the treatment of primary hyperhidrosis of the axilla.

ELIGIBILITY:
Inclusion Criteria:

* A healthy non-smoking male or female between 18-56 years of age
* Understand/accept obligation not to receive any other procedures in anatomical areas exhibiting axillary hyperhidrosis through 3 months prior to treatment
* Understand and accept the obligation and is logistically able to present for all scheduled follow-up visits
* Clinically diagnosed for primary hyperhidrosis of the axilla.
* A self assessed Hyperhidrosis Disease Severity Scale (HDSS) score of three (3) or four (4)

Exclusion Criteria:

* Clinical diagnosis of secondary hyperhidrosis
* Uncontrolled systemic disease
* Concurrent use of any hyperhidrosis treatments other than over the counter antiperspirants or deodorants
* Receipt of Botox or Dysport within the past six months
* Patients who refuse to stop using over the counter antiperspirants 24 hours prior to the day of surgery and each of the follow-up visits at 3 months and 6 months that Minors starch iodine tests may be performed.
* Patients using or having used within 7 days of baseline visit: cholinomimetic agents, anticholinergic agents, prescription antiperspirants, any herbal medicine treatments or any other treatments for hyperhidrosis except over the counter antiperspirant or planning to use such agents during the course of the study.
* Any previous liposuction/liposculpture or any type of surgery for hyperhidrosis; OR any other types of treatments for hyperhidrosis in the area to be treated in the past 6 months or planning to have any treatments for hyperhidrosis or surgery within the treatment area during the course of the study.
* Allergies to medication or local anesthesia required for the procedure
* A history of thrombophlebitis
* A history of acute infections
* A history of heart failure
* Received or is anticipated to receive antiplatelets, anticoagulants, thrombolytics, vitamin E or anti inflammatories within 2 weeks pre treatment
* An intolerance to anesthesia
* Any medical condition, that, in the investigator's opinion would interfere with the patient's participation in the study
* Taking medications that are photosensitive
* A history of keloid formation
* Is pregnant or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the course of the study
* Study subjects that can not maintain their pre-study exercise and diet routine over the course of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-06; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Krantz, Study Director — Cynosure, Inc.
Locations (1):
- Juva Skin and Laser Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nd:YAG Laser: Nd:YAG 1440nm Laser
  Nd:YAG Multiwavelength Diode Laser Using 1440nm Wavelength. A Rep Rate of 25 Hz was used.
  Each subject received 1 treatment using this laser.
Period: Overall Study
Arm/Group | Nd:YAG Laser
Started | 19
Completed | 17
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Nd:YAG Laser
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Asian | 1
  Race/Ethnicity: African American | 2
  Race/Ethnicity: African American/Caucasian | 1
  Race/Ethnicity: Hispanic | 0
  Race/Ethnicity: Caucasian | 15
Fitzpatrick Skin Score [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is.
  The scale comes from this source:
  Gupta, Sharma. Skin typing: Fitzpatrick grading and others. Clinics in Dermatology. 2019;37(5):430-436. doi:10.1016/j.clindermatol.2019.07.010
  Participants
    Fitzpatrick Skin Type I | 2
    Fitzpatrick Skin Type II | 8
    Fitzpatrick Skin Type III | 7
    Fitzpatrick Skin Type IV | 1
    Fitzpatrick Skin Type V | 1
    Fitzpatrick Skin Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Photographs Identified Accurately
Description: 3 trained blinded evaluators were asked to pick the post treatment photo from pre and post treatment photograph sets.
Time Frame: 3 Month Follow Up
Population: The subject was lost to follow up (not due to adverse events).
Measure: Mean (Standard Deviation); unit: % of photographs identified correctly
Arm/Group | Nd:YAG Laser
Number analyzed (Participants) | 18
% of photographs identified correctly | 84.8 (5.9)

2. Primary Outcome: Percentage of Photographs Identified Accurately
Description: 3 trained blinded evaluators were asked to pick the post treatment photo from pre and post treatment photograph sets.
Time Frame: 6 Month Follow Up
Population: Anything beyond the 3 month follow up was not required, and the subject chose not to come in.
Measure: Mean (Standard Deviation); unit: % of photographs identified correctly
Arm/Group | Nd:YAG Laser
Number analyzed (Participants) | 17
% of photographs identified correctly | 87.2 (12.3)

3. Secondary Outcome: Number of Participants With Changed and Unchanged Glands on Biopsy Sampling
Description: Hematoxylin and eosin (H&E) staining was performed on all pre and post treatment biopsy samples and evaluated by a pathologist to determine if there was any change in the subjects' glands at baseline vs. post last treatment. Changes in glands are characterized by reduction in quantity and size, in addition to changes in shape.
Time Frame: up to 3 months post last treatment
Population: The biopsy portion of the study was optional, so there were only 5 subjects.
Measure: Count of Participants; unit: Participants
Arm/Group | Nd:YAG Laser
Number analyzed (Participants) | 5
Participants
  # of Participants with Only Unchanged Glands | 3
  # of Participants with Changed Glands | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the study duration, around 12 months.
Arm/Group | Nd:YAG Laser
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 19/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nd:YAG Laser (N=19)
Numbness (Nervous system disorders) | 18
Pain (Nervous system disorders) | 19
Redness (Skin and subcutaneous tissue disorders) | 18
Swelling (Skin and subcutaneous tissue disorders) | 18
Bruising (Skin and subcutaneous tissue disorders) | 19
Itching (Skin and subcutaneous tissue disorders) | 15
Nodule (Skin and subcutaneous tissue disorders) | 0
Blister (Skin and subcutaneous tissue disorders) | 1
Hardness (Skin and subcutaneous tissue disorders) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.